CLINICAL TRIAL: NCT00842010
Title: Hyperglycemic Non Diabetic (HND) Hospital Patients: Are They Different From Diabetic Hyperglycemic and Non-Hyperglycemic Non-Diabetic(NHND) Patients?
Brief Title: Characteristics of Non Diabetic Hyperglycemic Inpatients
Status: Completed | Type: Observational
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Yannis Guerra, MD, Cook County Health
Other Study IDs: 06-063
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Inpatient; Hospital; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hyperglycemic without previous DM diagnosis: Patients with hyperglycemia, without previous diagnosis of diabetes
- Previous diagnosis of DM: Patients that have previous diagnosis of Diabetes Mellitus
- No previous DM diagnosis and no hyperglycemia: Patient with NO previous diagnosis of diabetes, and no hyperglycemia

SUMMARY:
Retrospective nested non-matched case control study comparing patients by glycemic status

DETAILED DESCRIPTION:
This retrospective nested non-matched case control study compared patients directly admitted to the General Medicine Wards, not transferred from ICU with

* hyperglycemia on admission but no previous diagnosis of diabetes
* diabetic hyperglycemic patients
* non hyperglycemic non diabetic patients from the same nested population.

The investigators' hypothesis is that the clinical characteristics and endpoints of the non diabetic hyperglycemics should be similar to the diabetic population and different from the non diabetic non hyperglycemic population.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to John H. Stroger Jr. Hospital
* Admitted to Internal Medicine Service from March-April 2006 and in October 2007

Exclusion Criteria:

* Transfer from any intensive care unit (medical or surgical)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nested sample obtained from patients admitted to John H. Stroger Jr. Hospital from March-April 2006 and in October 2007.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Length of stay | Measured 24 hours after patient is discharged. From day 1 of admission until day of discharge
  Hospital stay measured in days
Inpatient Mortality | From day 1 of admission until day of discharge
  Mortality measured in number of events

SECONDARY OUTCOMES:
Frequency of SIRS on admission | Measures obtained 24 hours after patient is discharged. Clinical data obtained on day 1 of admission
  Number of SIRS
Frequency of inpatient infection | From day 1 of admission until day of discharge
  Measured in number of events
Rate of use of intravenous glucose drip | From day 1 of admission until day of discharge
  Rate of use
Frequency of steroid use | From day 1 of admission until day of discharge
  Frequency of use

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Lacuesta, MD, Principal Investigator — John H. Stroger Jr. Hospital; Jyothsna Palla, MD, Study Chair — John H. Stroger Jr. Hospital; Yannis Guerra, MD, Study Chair — Rush University Hospital, John H. Stroger Jr. Hospital
Locations (1):
- John H. Stroger Jr. Hospital, Chicago, Illinois, United States